CLINICAL TRIAL: NCT01470352
Title: Multiparametric MRI Study of Endogenous Analgesia and Prediction the Efficacy of Migraine Pharmacological Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: d_yarnitsky (Other)
Responsible Party: Sponsor-Investigator, d_yarnitsky, Head of Neurology Department, Rambam Health Care Campus
Organization: Rambam Health Care Campus (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Migrain-0265-11CTIL
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Migraine
Keywords: migraine; pain; CPM; offset analgesia; fMRI
MeSH Terms: conditions — Migraine Disorders; Pain | interventions — Duloxetine Hydrochloride; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Doluxetine; Drug: Placebo
- treatment (Active Comparator): Duloxetine will be given in a daily dose of 30 mg for 5 weeks
  Interventions: Drug: Doluxetine; Drug: Placebo

INTERVENTIONS:
Drug: Doluxetine — 30 mg/d
  Other Names: duloxetine
Drug: Placebo — suger pill 30mg/d
  Other Names: sugar

SUMMARY:
To delineate brain mechanisms that subserve EA in the healthy state and to identify alterations in mechanisms supporting EA in chronic pain and their therapeutic relevance. Individuals with migraine will be examined between episodes in order to assess basal alterations in the efficiency of spatial and temporal filtering of noxious information. This population provides the unique opportunity to examine such processes without confounds arising from ongoing pain.

DETAILED DESCRIPTION:
Pain is a uniquely individual experience that is powerfully shaped by the action of descending control mechanisms. These systems may play crucial roles in the moment-to-moment tuning of the sensitivity, spatial, and temporal response characteristics of nociceptive processing mechanisms during both acute and pathological pain states. However, these systems remain poorly understood in human subjects. The proposed research will use psychophysics and multiparametric MRI to (i) delineate the brain mechanisms that subserve and regulate endogenous analgesia (EA) in the healthy state and (ii) to identify alterations in mechanisms supporting EA in chronic pain and their therapeutic relevance. In both healthy subjects and chronic pain patients, EA will be probed using the DNIC (diffuse noxious inhibitory controls) and offset analgesia paradigms. Functional MRI will examine activation of brainstem mechanisms important in EA, while both functional and structural connectivity analyses will assess the regulation of these brainstem mechanisms by cerebral cortical regions involved in attention and affect. One pathological painful condition, migraine, will be examined since it allows changes in EA associated with chronic pain to be investigated between episodes of pain. Finally, EA and EA associated structural and functional parameters will be used to predict the efficacy of one compound, amitriptyline, to treat migraine in individual patients. Taken together, the proposed research will provide substantial insights into basic mechanisms supporting and regulating EA and can provide a foundation for mechanism-based individualized choice of therapy that may benefit all chronic pain patients.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with migraine based on the International Headache Society (IHS) criteria 1 that have >4 attacks/month, both with and without aura

Exclusion Criteria:

* patients receiving any migraine preventive treatment during last 3 months or prior treatment with amytriptiline
* other chronic pain conditions
* psychiatric, other neurological diseases, language barrier or cognitive dysfunction

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 179 (Actual)
Dates: Start 2011-11-16 (Actual); Primary Completion 2017-11-06 (Actual); Study Completion 2017-11-06 (Actual)

PRIMARY OUTCOMES:
Therapeutic response to the analgesic drugs | 2 month
  The level of pain relief

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam health care campus, Haifa, Israel